CLINICAL TRIAL: NCT02748694
Title: A Randomized, Double -Blind, Placebo-Controlled, Phase 1, Ascending Oral Single and Multiple Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAK-041 in Healthy Subjects and Subjects With Stable Schizophrenia and a Randomized Open-Label, Single Dose, Parallel Design to Evaluate the Relative Bioavailability and Effect of Food on the Pharmacokinetics of TAK-041 Tablet Formulation in Healthy Subjects
Brief Title: Phase 1 TAK-041 First-in-Human Safety, Tolerability, and Pharmacokinetics Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TAK-041-1001; U1111-1178-6559 (Registry Identifier: WHO)
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers; Schizophrenia
Keywords: Drug Therapy
MeSH Terms: conditions — Schizophrenia | interventions — TAK-041

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Part 1 (SRD): Placebo Cohorts 1-5 (Placebo Comparator): TAK-041 placebo-matching suspension, orally, once on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-041 Placebo
- Part 1 (SRD): Cohort 1: TAK-041 5/20 mg (Experimental): TAK-041 5 mg, suspension, orally, once on Day 1 in fasted healthy participants in the SRD period. Participants also received 20 mg, suspension, orally, once on Day 8 in the SRD period.
  Interventions: Drug: TAK-041
- Part 1 (SRD): Cohort 2: TAK-041 10/40 mg (Experimental): TAK-041 10 mg, suspension, orally, once on Day 1 in fasted healthy participants in the SRD period. Participants also received 40 mg, suspension, orally, once on Day 8 in the SRD period.
  Interventions: Drug: TAK-041
- Part 1 (SRD): Cohort 3: TAK-041 80 mg (Experimental): TAK-041 80 mg, suspension, orally, once on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-041
- Part 1 (SRD): Cohort 4: TAK-041 120 mg (Experimental): TAK-041 120 mg, suspension, orally, once on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-041
- Part 1 (SRD): Cohort 5: TAK-041 160 mg (Experimental): TAK-041 160 mg, suspension, orally, once on Day 1 in fasted healthy participants in the SRD period.
  Interventions: Drug: TAK-041
- Part 2 (MRD): Placebo Cohorts 1-4 (Placebo Comparator): TAK-041 placebo-matching suspension, orally, once on Day 1 in fasted healthy participants in the multiple-rising dose (MRD) period.
  Interventions: Drug: TAK-041 Placebo
- Part 2 (MRD): Cohort 1: TAK-041 40/20 mg (Experimental): TAK-041 40 mg as loading dose, suspension, orally, once on Day 1 in fasted healthy participants followed by 20 mg (half the initial dose) as a maintenance dose on Days 8, 15 and 22 in the MRD period.
  Interventions: Drug: TAK-041
- Part 2 (MRD): Cohort 2: TAK-041 80/40 mg (Experimental): TAK-041 80 mg as loading dose, suspension, orally, once on Day 1 in fasted healthy participants followed by 40 mg (half the initial dose) as a maintenance dose on Days 8, 15 and 22 in the MRD period.
  Interventions: Drug: TAK-041
- Part 2 (MRD): Cohort 3: TAK-041 120/60 mg (Experimental): TAK-041 120 mg as loading dose, suspension, orally, once on Day 1 in fasted healthy participants followed by 60 mg (half the initial dose) as a maintenance dose on Days 8, 15 and 22 in the MRD period.
  Interventions: Drug: TAK-041
- Part 2 (MRD): Cohort 4: TAK-041 160/80 mg (Experimental): TAK-041 160 mg as loading dose, suspension, orally, once on Day 1 in fasted healthy participants followed by 80 mg (half the initial dose) as a maintenance dose on Days 8, 15 and 22 in the MRD period.
  Interventions: Drug: TAK-041
- Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A (Experimental): TAK-041 40 mg, tablet, orally, once on Day 1 in fasted state (Regimen A) in Cohort 1.
  Interventions: Drug: TAK-041
- Part 3: RBA/Food Effect: Regimen B (Experimental): TAK-041 40 mg, tablet, orally, once on Day 1 in fed state (Regimen B) in Cohort 2.
  Interventions: Drug: TAK-041
- Part 4: MRD: Placebo (Placebo Comparator): TAK-041 placebo-matching, suspension, orally, on Days 1, 8, 15 and 22 in participants with schizophrenia
  Interventions: Drug: TAK-041; Drug: TAK-041 Placebo
- Part 4: MRD: TAK-041 160/80 mg (Experimental): TAK-041 160 mg as loading dose, suspension, orally, once on Day 1 followed by 80 mg (half the initial dose) as a maintenance dose on Days 8, 15 and 22 in participants with schizophrenia.
  Interventions: Drug: TAK-041

INTERVENTIONS:
Drug: TAK-041 — TAK-041 tablets or oral suspension.
  Arms: Part 1 (SRD): Cohort 1: TAK-041 5/20 mg; Part 1 (SRD): Cohort 2: TAK-041 10/40 mg; Part 1 (SRD): Cohort 3: TAK-041 80 mg; Part 1 (SRD): Cohort 4: TAK-041 120 mg; Part 1 (SRD): Cohort 5: TAK-041 160 mg; Part 2 (MRD): Cohort 1: TAK-041 40/20 mg; Part 2 (MRD): Cohort 2: TAK-041 80/40 mg; Part 2 (MRD): Cohort 3: TAK-041 120/60 mg; Part 2 (MRD): Cohort 4: TAK-041 160/80 mg; Part 3: RBA/Food Effect: Regimen B; Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A; Part 4: MRD: Placebo; Part 4: MRD: TAK-041 160/80 mg
Drug: TAK-041 Placebo — TAK-041 placebo-matching suspension or tablet.
  Arms: Part 1 (SRD): Placebo Cohorts 1-5; Part 2 (MRD): Placebo Cohorts 1-4; Part 4: MRD: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of TAK-041:

1. Following oral single and multiple doses in healthy participants.
2. As add-on therapy to antipsychotics in stable schizophrenia participants.
3. To determine the oral bioavailability of the TAK-041 tablet formulation compared to the oral suspension formulation in the fasted state.
4. To assess the effect of food on the PK of TAK-041 in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-041. TAK-041 is being tested to evaluate its safety, tolerability, and PK of single and multiple doses in healthy participants and as add-on therapy to antipsychotics in participants with stable schizophrenia. This study will also assess the oral bioavailability in healthy participants administered with tablet formulation compared to oral suspension formulation in fasted state, and effect of high-fat, high-calorie meal on the PK of single dose of TAK-041 tablet formulation.

The study will enroll approximately 114 participants. The study is composed of 4 parts. Part 1 (single-rising dose [SRD], alternating panel design and a sequential panel design), Part 2 (multiple-rising dose [MRD], sequential panel design), Part 3 (open label parallel design), and Part 4 (single dose cohort).

Part 1 consists of 5 cohorts, participants in Cohorts 1 and 2 will be randomly assigned (by chance, like flipping a coin) to treatment sequences of 2 periods and for Cohorts 3 to 5 participants will be assigned to a single dose sequential-panel:

* TAK-041 5-160 mg
* Placebo (inactive) - this is a similar formulation that looks like the study drug but has no active ingredient.

Part 2 consists of 4 cohorts, participants will be randomly assigned to one of the two treatments:

* TAK-041
* Placebo Dose levels for Part 2 cohort 1 will be based on emerging safety/tolerability and PK data from Part 1. The dose levels for Part 2 Cohorts 2 onwards will be based on emerging safety/tolerability and available PK data from Part 1 and from preceding cohorts in Part 2.

Part 3 consists of 2 cohorts, participants will be randomly assigned to one of the two treatments under fasted state or fed state:

* TAK-041 40 mg tablet (Fasted state)
* TAK-041 40 mg tablet (Fed state)

Part 4 consists of 1 cohort, participants will be randomly assigned to one of the two treatments:

* TAK-041
* Placebo The dose levels for Part 4 will be based upon the emerging safety/tolerability and PK data of same dose in healthy participants from Part 2.

This single center trial will be conducted in the United States. Participants will remain confined to the study site from check-in (Day -1) through Days 5 of each period in Part 1, on Days -2 to 3, Days 7 to 10, Days 14 to 17, Day 21 to 24 in Part 2, on Days 1 to 3 in Part 3, and on Days -2 to 3, Days 7 to 10, Days 14 to 17, Days 21 to 24 in Part 4. A final visit that completes the study will occur 12 to 16 days after the last safety and PK follow-up visit in Part 1, 2 and 4, and 18 days after dosing in Part 3.

ELIGIBILITY:
Inclusion Criteria:

Healthy Participants and Participants with Schizophrenia:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any participant procedures including requesting that a participant fast for any laboratory evaluations.
3. The participant is willing to comply with study restrictions described in the protocol.
4. The participant is a healthy adult man or woman (of non-childbearing potential as described in the protocol)
5. The participant is aged 18 to 55 years, inclusive, at the time of informed consent.
6. The participant weighs at least 45 kilogram (kg) (99 pound [lb]) with a body mass index from 18 to 32 kilogram per square meter (kg/m^2) for healthy participants and up to 40.5 kg/m^2 for participants with schizophrenia, inclusive at screening.
7. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception (as defined in the protocol)from signing of informed consent throughout the duration of the study and for 145 days have elapsed since the last dose of study drug.

Participants with schizophrenia only-:

1. Is on a stable dose of an antipsychotic medication for at least 2 months as documented by medical history and assessed by site staff.
2. Meets schizophrenia criteria as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) by the Mini International Neuropsychiatric Interview (MINI).
3. Has Positive and Negative Syndrome Scale (PANSS) total score less than or equal to (<=) 90 and PANSS Negative Symptom Factor Score (NSFS; Sum of PANSS N1, N2, N3, N4, N6, G7, and G16) greater than or equal to (>=) 15 at screening and baseline (Day-1).
4. Has stable screening and baseline (Day -1) PANSS and NSFS total scores (less than [<] 20 percent (%) change).

Exclusion Criteria:

Healthy Participants:

1. The participant has received any investigational compound within 30 days prior to the first dose of study drug, or due to the half-life of the investigational drug is likely to still have detectable plasma levels of that compound.
2. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (example spouse, parent, child, sibling) or may consent under duress
3. The participant has a known hypersensitivity to any component of the formulation of TAK-041.
4. The participant has a positive urine/blood drug result for drugs of abuse (defined as any illicit drug use) at Screening or Check-in (Day -1).
5. The participant taken any excluded medication, supplements, or food products during the time periods listed in the protocol.
6. The participant is lactose intolerant (Part3 only).
7. If female, the participant is of childbearing potential (example, premenopausal, not sterilized).
8. If male, the participant intends to donate sperm during the course of this study or for 145 days have elapsed since the last dose of study drug.
9. The participant has evidence of current active cardiovascular, central nervous system, hepatobiliary disease including history of biliary tree disorders, gallstones, endoscopic retrograde cholangio pancreatography (ERCP), and/or cholecystectomy, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma, hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory test results (including elevated alkaline phosphatase (ALP), elevated bilirubin, elevated GGT, or elevated 5'-nucleotidase) that in the judgment of the principal investigator represents a reasonable suspicion of a disease that would contraindicate taking TAK-041, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, cholestasis, seizure disorders, and cardiac arrhythmias.
10. The participant has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (that is, a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention).
11. Had major surgery, or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to Screening.
12. The participant has a history of cancer, except basal cell carcinoma that has been in remission for at least 5 years prior to Day 1. Participant has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody at Screening or a known history of human immunodeficiency virus (HIV) infection.
13. The participant has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 21 days prior to Check-in on Day -1. Cotinine test is positive at Screening or Day -1.
14. The participant has poor peripheral venous access.
15. Had a transfusion of any blood product within 30 days prior to Day 1.
16. Participant has a Screening or Check-in abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature of the principal investigator or a medically qualified sub-investigator.
17. The participant has a sustained resting heart rate outside the range 40 to 100 beats per minute (bpm), confirmed on repeat testing within a maximum of 30 minutes, at Screening or Check-in.
18. The participant has a QT interval with Fridericia correction method (QTcF) >450 millisecond (ms) or PR outside the range 120 to 220 ms, confirmed on repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in.
19. The participant has abnormal Screening or Check-in laboratory values (> upper limit of normal [ULN] for the respective serum chemistries) of alanine transaminase (ALT), aspartate aminotransferase (AST), total bilirubin (TBILI), ALP, gamma-glutamyl transpeptidase (GGT), 5'nucleotidase (Screening only) and/or abnormal urine osmolality, confirmed upon repeat testing.
20. The participant has a clinically significant history of head injury or trauma associated with loss of consciousness for >15 minutes.
21. Is considered by the investigator to be at an imminent risk of suicide injury to self, other, property, or participants who within the past year prior to Screening have attempted suicide. Participants having positive answer on item 4 or 5 on Columbia Suicide Severity Rating Scale (C-SSRS) (based on the past year) prior to randomization are excluded.
22. The participant has a history of significant skin reactions (hypersensitivity) to adhesives, metals or plastic; this criterion applies only to participants participating in the study of the two wearable digital devices.

Participants with schizophrenia only:

1. Has an undetectable level of baseline antipsychotic medication at Screening.
2. Has a lifetime diagnosis of schizoaffective disorder; a lifetime diagnosis of bipolar disorder; or a lifetime diagnosis of obsessive compulsive disorder based on the Mini International Neuropsychiatric Interview (MINI) combined with the general psychiatric evaluation. As an exception, participants with a historical prior lifetime diagnosis of schizoaffective disorder may be enrolled in the study with sponsor or designee approval provided that the principal investigator can attest that the participant's overall history and current clinical presentation and history is most consistent with schizophrenia, not schizoaffective disorder.
3. Has a recent (within the last 6 months) diagnosis of panic disorder, depressive episode, or other comorbid psychiatric conditions requiring clinical attention based on the MINI for DSM-5 and the general psychiatric evaluation.
4. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as 4 or more alcoholic beverages per day) within 1 year prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
5. Has a diagnosis of substance use disorder (with the exception of nicotine dependence) within the preceding 6 months based on the MINI for DSM-5 and the general psychiatric evaluation.
6. Has evidence or history of current clinically significant cardiovascular disease, including uncontrolled hypertension (standing or supine diastolic blood pressure >90 millimeter of mercury (mm Hg) and/or standing or supine systolic blood pressure >145 mm Hg, with or without treatment), symptomatic ischemic heart disease, uncompensated heart failure or recent (past 12 months) acute myocardial infarction or bypass surgery. Controlled essential hypertension, non-clinically significant sinus bradycardia and sinus tachycardia will not be considered significant medical illnesses and would not exclude a participant from the study. Other well-controlled medical illnesses may be permitted that do not increase hepatic risks or other safety risks to the participant's participation in the judgement of the investigator in consultation with the sponsor or designee.
7. Has evidence of clinically significant extrapyramidal symptoms as measured by a Simson-Angus Scale (SAS) score >6.
8. The participant has evidence of depression as measured by a Calgary Depression Score (CDSS) score >9.
9. Has received TAK-041 in a previous clinical study; or has previously or is currently participating in this study; has received treatment with other experimental therapies within the preceding 60 days or <5 half-lives prior to randomization, whichever is longer; has participated in 2 or more clinical studies within 12 months prior to Screening; or has participated in a clinical study for a psychiatric condition that is exclusionary per this protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2019-09-22 (Actual); Study Completion 2019-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Parexel Early Phase Clinic Unit- Los Angeles, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Yin W, Han D, Khudyakov P, Behrje R, Posener J, Laurenza A, Arkilo D. A phase 1 study to evaluate the safety, tolerability and pharmacokinetics of TAK-041 in healthy participants and patients with stable schizophrenia. Br J Clin Pharmacol. 2022 Aug;88(8):3872-3882. doi: 10.1111/bcp.15305. Epub 2022 Apr 17. PMID 35277995

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in the United States from 09 May 2016 to 22 September 2019.
Pre-assignment Details: Healthy participants were enrolled in Parts 1 to 3 to receive TAK-041 or placebo in this study as a single-rising dose (SRD), multiple-rising dose (MRD) or to assess the effect of food on drug's bioavailability. Participants with stable schizophrenia received TAK-041 or placebo as an add-on therapy in Part 4.
Groups:
- Part 1 (SRD): Placebo Cohorts 1-5: TAK-041 placebo-matching suspension, orally, once on Day 1 in fasted healthy participants in the single-rising dose (SRD) period.
Period: Overall Study
Arm/Group | Part 1 (SRD): Placebo Cohorts 1-5 | Part 1 (SRD): Cohort 1: TAK-041 5/20 mg | Part 1 (SRD): Cohort 2: TAK-041 10/40 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg | Part 2 (MRD): Placebo Cohorts 1-4 | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part 4: MRD: Placebo | Part 4: MRD: TAK-041 160/80 mg
Started | 10 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 9 | 9 | 8 | 16
Completed | 10 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 9 | 9 | 8 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Voluntary Withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Part 2 (MRD): Placebo Cohorts 1-4: TAK-041 placebo-matching suspension, orally, once on Day 1 in fasted healthy participants in the MRD period.
- Total: Total of all reporting groups
Arm/Group | Part 1 (SRD): Placebo Cohorts 1-5 | Part 1 (SRD): Cohort 1: TAK-041 5/20 mg | Part 1 (SRD): Cohort 2: TAK-041 10/40 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg | Part 2 (MRD): Placebo Cohorts 1-4 | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part 4: MRD: Placebo | Part 4: MRD: TAK-041 160/80 mg | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 9 | 9 | 8 | 16 | 114
Age, Continuous [Mean (Full Range); unit: years] | 40.6 [26 to 53] | 36.8 [27 to 54] | 29.3 [22 to 38] | 44.2 [37 to 52] | 42.3 [33 to 52] | 40.5 [25 to 54] | 35.5 [25 to 50] | 39.5 [26 to 55] | 38.3 [23 to 55] | 37.7 [27 to 49] | 42.5 [30 to 53] | 35.6 [23 to 51] | 34.1 [26 to 54] | 45.8 [34 to 55] | 44.3 [28 to 53] | 39.46 [22 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 2 | 1 | 2 | 3 | 24
  Male | 8 | 5 | 4 | 4 | 4 | 5 | 7 | 4 | 5 | 5 | 5 | 7 | 8 | 6 | 13 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 2 | 0 | 3 | 2 | 1 | 0 | 2 | 1 | 2 | 2 | 1 | 1 | 1 | 22
  Not Hispanic or Latino | 6 | 6 | 4 | 6 | 3 | 4 | 7 | 6 | 4 | 5 | 4 | 7 | 8 | 7 | 15 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 0 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 2 | 2 | 3 | 0 | 4 | 3 | 2 | 1 | 1 | 0 | 1 | 2 | 5 | 8 | 35
  White | 7 | 2 | 1 | 3 | 5 | 2 | 5 | 2 | 3 | 4 | 5 | 8 | 4 | 3 | 5 | 59
  More than one race | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 9 | 9 | 8 | 16 | 114
Height [Mean (Full Range); unit: cm] | 176.9 [162 to 190] | 174.3 [162 to 184] | 171.2 [157 to 185] | 175.2 [162 to 185] | 164.8 [151 to 178] | 178.3 [164 to 190] | 178.3 [169 to 185] | 174.2 [168 to 180] | 168.3 [151 to 176] | 173.8 [160 to 184] | 173.0 [159 to 184] | 175.3 [163 to 189] | 175.7 [168 to 191] | 173.9 [153 to 183] | 174.9 [157 to 191] | 174.24 [151 to 191]
Weight [Mean (Full Range); unit: kg] | 79.68 [60.8 to 105.0] | 78.63 [62.9 to 99.0] | 74.43 [65.7 to 83.6] | 86.97 [76.3 to 103.4] | 68.52 [57.7 to 77.5] | 89.83 [79.0 to 105.8] | 81.79 [73.5 to 92.2] | 83.40 [60.5 to 99.8] | 77.20 [54.8 to 90.9] | 78.22 [62.5 to 104.0] | 76.43 [64.3 to 92.5] | 76.07 [63.2 to 84.9] | 79.42 [56.7 to 94.3] | 91.46 [71.2 to 131.1] | 98.58 [66.5 to 129.5] | 81.82 [54.8 to 131.1]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] — BMI = Weight(kg)/height(m)^2.
  kg/m^2 | 25.47 [19.7 to 31.0] | 25.91 [19.6 to 30.9] | 25.43 [23.7 to 26.7] | 28.36 [23.3 to 31.5] | 25.28 [21.3 to 27.5] | 28.22 [25.9 to 31.0] | 25.80 [22.0 to 30.3] | 27.63 [18.9 to 31.9] | 27.14 [20.1 to 29.4] | 25.74 [21.6 to 31.4] | 25.44 [22.2 to 29.4] | 24.76 [21.2 to 28.7] | 25.68 [19.4 to 31.5] | 30.31 [21.7 to 39.6] | 32.05 [21.6 to 39.1] | 27.24 [18.9 to 39.6]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug or due to a study procedure; it did not necessarily have to have a causal relationship with this treatment. A TEAE was defined as an AE that occurred or worsened after receiving the first dose of study drug and within 6 weeks after the last dose of study drug. A TEAE may also have been a pre-treatment AE or a concurrent medical condition diagnosed before the date of first dose of study drug that increased in severity after the start of dosing.
Time Frame: From the first dose of study drug up to 42 days after the last dose of study drug (Up to 12 weeks)
Population: Safety Set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Part 1 (SRD): Cohort 1: TAK-041 5 mg: TAK-041 5 mg, suspension, orally, once on Day 1 in fasted healthy participants in the SRD period.
- Part 1 (SRD): Cohort 2: TAK-041 10 mg: TAK-041 10 mg, suspension, orally, once on Day 1 in fasted healthy participants in the SRD period.
- Part 1 (SRD): Cohort 1: TAK-041 20 mg: TAK-041 20 mg, suspension, orally, once on Day 8 in the SRD period.
- Part 1 (SRD): Cohort 2: TAK-041 40 mg: TAK-041 40 mg, suspension, orally, once on Day 8 in the SRD period.
Arm/Group | Part 1 (SRD): Placebo Cohorts 1-5 | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg | Part 2 (MRD): Placebo Cohorts 1-4 | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part 4: MRD: Placebo | Part 4: MRD: TAK-041 160/80 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 9 | 9 | 8 | 16
percentage of participants | 40.0 | 0 | 0 | 0 | 0 | 33.3 | 33.3 | 33.3 | 37.5 | 66.7 | 66.7 | 50.0 | 83.3 | 11.1 | 22.2 | 75.0 | 56.3

2. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug or due to a study procedure; it did not necessarily have to have a causal relationship with this treatment.
Time Frame: From the first dose of study drug up to 42 days after the last dose of study drug (Up to 12 weeks)
Population: Safety Set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (SRD): Placebo Cohorts 1-5 | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg | Part 2 (MRD): Placebo Cohorts 1-4 | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part 4: MRD: Placebo | Part 4: MRD: TAK-041 160/80 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 9 | 9 | 8 | 16
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Markedly Abnormal Value (MAV) Criteria for Safety Laboratory Tests At Least Once Post-dose
Description: Clinical laboratory tests included serum chemistry, hematology and urinalysis. MAV criteria:Alanine aminotransferase(U/L) >3 x upper limit of normal(ULN);albumin<2.5g/dL,<25g/L;alkaline phosphatase (U/L)>3 x ULN; aspartate aminotransferase (U/L)>3 x ULN;bicarbonate<8.0 mmol/L; bilirubin>2.0mg/dL, >34.2 μmol/L;blood urea nitrogen>30 mg/dL,>10.7mmol/L;calcium<7.0 mg/dL,<1.75 mmol/L, >11.5 mg/dL,>2.88 mmol/L;chloride<75 mmol/L,>126 mmol/L;creatine kinase(U/L) >5 xULN; creatinine>2.0 mg/dL,>177μmol/L;direct bilirubin>2 x ULN;gamma glutamyl transferase (U/L)>3 x ULN;glucose<50 mg/dL,<2.8 mmol/L,>350 mg/dL,>19.4 mmol/L;potassium<3.0 mmol/L >6.0 mmol/L; protein(g/L)<0.8 x LLN >1.2 x ULN;sodium<130mmol/L >150mmol/L;erythrocytes(10^12erythrocytes/L) <0.8 x LLN,>1.2 x ULN;hematocrit(fraction of 1)<0.8 x LLN,>1.2xULN;hemoglobin(g/L)<0.8 x LLN>1.2 x ULN;leukocytes(10^9 leukocytes/L)<0.5 x LLN >1.5 x ULN;platelets(10^9 platelets/L)<75->600. Categories with at least one participant are reported.
Time Frame: From the first dose of study drug up to 42 days after the last dose of study drug (Up to 12 weeks)
Population: Safety Set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (SRD): Placebo Cohorts 1-5 | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg | Part 2 (MRD): Placebo Cohorts 1-4 | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part 4: MRD: Placebo | Part 4: MRD: TAK-041 160/80 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 9 | 9 | 8 | 16
percentage of participants
  Creatine Kinase, > 5 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 12.5 | 0 | 0 | 0 | 0 | 0 | 11.1 | 0 | 12.5
  Glucose < 50 mg/dL, < 2.8 mmol/L | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase, > 3 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11.1 | 0 | 6.3
  Leukocytes, > 1.5 x ULN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6.3
  Platelets, > 600 10^9 platelets/L | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6.3

4. Primary Outcome: Percentage of Participants With Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post-dose
Description: Vital signs included oral body temperature measurement, supine and standing blood pressure, respiration rate, and pulse. Pulse and blood pressure was measured after 5 minutes supine and again at 1 and 3 minutes after standing. The markedly abnormal value (MAV) criteria for vital signs included systolic blood pressure < 85 mmHg, > 180 mmHg; diastolic blood pressure < 50 mmHg, > 110 mmHg; pulse < 50 beats/min, > 120 beats/min; temperature < 35.6 C > 37.7 C. Categories with data in at least one arm group are reported.
Time Frame: From the first dose of study drug up to 42 days after the last dose of study drug (Up to 12 weeks)
Population: Safety Set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (SRD): Placebo Cohorts 1-5 | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg | Part 2 (MRD): Placebo Cohorts 1-4 | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part 4: MRD: Placebo | Part 4: MRD: TAK-041 160/80 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 9 | 9 | 8 | 16
percentage of participants
  Systolic Blood Pressure, Standing, < 85 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5 | 0
  Systolic Blood Pressure, Supine, < 85 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic Blood Pressure, 5 min Supine, < 85 mmHg | 10.0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5 | 6.3
  Systolic Blood Pressure, 1 min Standing, < 85 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 12.5 | 0
  Systolic Blood Pressure, 3 min Standing, < 85 mmHg | 10.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5 | 0
  Diastolic Blood Pressure, 5 min Supine, < 50 mmHg | 10.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 11.1 | 0 | 0
  Diastolic Blood Pressure,1 min Standing,>110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6.3
  Diastolic Blood Pressure,3 min Standing,>110 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12.5 | 6.3
  Pulse Rate, Standing, < 50 beats/min | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0
  Pulse Rate, Standing, > 120 beats/min | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 6.3
  Pulse Rate, Supine, < 50 beats/min | 10.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 12.5 | 0
  Pulse Rate, 5 min Supine, < 50 beats/min | 50.0 | 16.7 | 33.3 | 33.3 | 33.3 | 16.7 | 33.3 | 50.0 | 62.5 | 33.3 | 16.7 | 83.3 | 33.3 | 0 | 33.3 | 12.5 | 12.5
  Pulse Rate, 1 min Standing, < 50 beats/min | 10.0 | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 33.3 | 16.7 | 0 | 0 | 0 | 0
  Pulse Rate, 1 min Standing, > 120 beats/min | 0 | 0 | 0 | 0 | 16.7 | 0 | 16.7 | 0 | 0 | 0 | 33.3 | 0 | 0 | 0 | 0 | 25.0 | 12.5
  Pulse Rate, 3 min Standing, < 50 beats/min | 10.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33.3 | 0 | 0 | 0 | 0 | 0
  Pulse Rate, 3 min Standing, > 120 beats/min | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33.3 | 0 | 0 | 0 | 0 | 0 | 25.0 | 12.5
  Temperature, < 35.6 C | 20.0 | 0 | 0 | 0 | 0 | 33.3 | 16.7 | 33.3 | 37.5 | 33.3 | 16.7 | 16.7 | 33.3 | 11.1 | 0 | 25.0 | 31.3

5. Primary Outcome: Percentage of Participants With Markedly Abnormal Criteria for 12-Lead Electrocardiogram (ECG) Parameters at Least Once Post-dose
Description: The markedly abnormal value (MAV) criteria for 12-lead ECG parameters included ECG Mean Heart Rate < 50 beats/min, > 120 beats/min; PR Interval, Aggregate <= 80 msec, >= 200 msec; QRS Duration, Aggregate <= 80 msec, >= 180 msec; QTcB Interval, Aggregate <= 300 msec, >= 500 msec OR (>= 30 msec change from baseline and >= 450 msec); QTcF Interval, Aggregate <= 300 msec, >= 500 msec OR (>= 30 msec change from baseline and >= 450 msec). Categories with data in at least one arm group are reported.
Time Frame: From the first dose of study drug up to 42 days after the last dose of study drug (Up to 12 weeks)
Population: Safety Set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 (SRD): Placebo Cohorts 1-5 | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg | Part 2 (MRD): Placebo Cohorts 1-4 | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part 4: MRD: Placebo | Part 4: MRD: TAK-041 160/80 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 9 | 9 | 8 | 16
percentage of participants
  ECG Mean Heart Rate, < 50 beats/min | 20.0 | 16.7 | 33.3 | 50.0 | 33.3 | 0 | 16.7 | 50.0 | 37.5 | 16.7 | 16.7 | 66.7 | 33.3 | 0 | 22.2 | 12.5 | 12.5
  PR Interval, Aggregate, >= 200 msec | 0 | 33.3 | 33.3 | 33.3 | 33.3 | 16.7 | 16.7 | 0 | 25.0 | 0 | 0 | 0 | 0 | 0 | 11.1 | 12.5 | 12.5
  QTcB Interval, Aggregate, >= 500 msec | 10.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6.3
  QTcF Interval, Aggregate, >= 500 msec | 0 | 0 | 0 | 0 | 0 | 16.7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS Duration, Aggregate, <= 80 msec | 20.0 | 33.3 | 50.0 | 33.3 | 50.0 | 33.3 | 33.3 | 16.7 | 0 | 33.3 | 33.3 | 66.7 | 16.7 | 33.3 | 11.1 | 75.0 | 31.3

6. Primary Outcome: Part 2: Percentage of Participants Who Experienced Clinically Significant Abnormal Changes in Continuous 12-Lead Holter ECG Measurements at Least Once Post-Dose
Description: The markedly abnormal value (MAV) criteria for continuous 12-lead Holter ECG parameters included ECG Mean Heart Rate < 50 beats/min, > 120 beats/min; PR Interval, Aggregate <= 80 msec, >= 200 msec; QRS Duration, Aggregate <= 80 msec, >= 180 msec; QTcB Interval, Aggregate <= 300 msec, >= 500 msec OR (>= 30 msec change from baseline and >= 450 msec); QTcF Interval, Aggregate <= 300 msec, >= 500 msec OR (>= 30 msec change from baseline and >= 450 msec). Categories with data in at least one arm group are reported.
Time Frame: Part 2: from first dose up to Day 66
Population: Safety Set included all participants who were enrolled and received at least 1 dose of study drug. Continuous 12-lead Holter ECG monitoring was performed in Part 2 only.
Measure: Number; unit: percentage of participants
Arm/Group | Part 2 (MRD): Placebo Cohorts 1-4 | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
percentage of participants
  ECG Mean Heart Rate, < 50 beats/min | 0 | 0 | 0 | 50.0 | 16.7
  PR Interval, Aggregate, >= 200 msec | 25.0 | 0 | 0 | 0 | 0
  QRS Duration, Aggregate, <= 80 msec | 0 | 0 | 16.7 | 0 | 0

7. Primary Outcome: Part 3: Cmax: Maximum Observed Plasma Concentration for TAK-041 in RBA/Food Effect Participants [Day 1]
Time Frame: Part 3: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Population: Pharmacokinetic (PK) Set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in the urine. Data for Regimen C were combined from Part 1 Cohort 2 and Part 2 Cohort 1 (Day 1) to report RBA/food effect on suspension formulation.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Part3:RBA/Food Effect:Regimen C-Part 1 Cohort2,Part 2 Cohort 1: Regimen C included participants from Part 1 Cohort 2 and Part 2 Cohort 1 who received TAK-041, 40 mg suspension, orally on Day 1 in fasted condition.
Arm/Group | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part3:RBA/Food Effect:Regimen C-Part 1 Cohort2,Part 2 Cohort 1
Number analyzed (Participants) | 9 | 9 | 12
ng/mL | 715.4 (192.54) | 838.3 (176.04) | 648.4 (158.67)

8. Primary Outcome: Part 3: AUC96: Area Under the Plasma Concentration-Time Curve From Time 0 to 96 Hours (AUC96) for TAK-041 in RBA/Food Effect Participants [Day 1]
Time Frame: Part 3: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Population: PK Set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in the urine. Data for Regimen C were combined from Part 1 Cohort 2 and Part 2 Cohort 1 (Day 1) to report RBA/food effect on suspension formulation.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part3:RBA/Food Effect:Regimen C-Part 1 Cohort2,Part 2 Cohort 1
Number analyzed (Participants) | 9 | 9 | 12
h*ng/mL | 41564.5 (7713.08) | 45499.1 (16007.58) | 37795.2 (5667.55)

9. Secondary Outcome: Part 1: Cmax: Maximum Observed Plasma Concentration for TAK-041 in SRD Participants [Day 1]
Time Frame: Part 1: Day 1 pre-dose and at multiple time points post dose, up to 96 hours for Cohorts 1 and 2; up to 168 hours for Cohorts 3-5
Population: PK Set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in the urine.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL | 139.8 (15.25) | 193.3 (27.75) | 909.5 (225.29) | 1200.0 (147.38) | 1121.7 (175.31)

10. Secondary Outcome: Part 1: Cmax: Maximum Observed Plasma Concentration for TAK-041 in SRD Participants [Day 8], Cohorts 1 (20 mg) and 2 (40 mg) Only
Time Frame: Part 1: Pre-dose on Day 8 and at multiple timepoints (Up to 96 hours) post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg
Number analyzed (Participants) | 6 | 6
ng/mL | 450.5 (90.25) | 747.2 (103.22)

11. Secondary Outcome: Parts 2 and 4: Cmax: Maximum Observed Plasma Concentration for TAK-041 in MRD Participants [Day 1]
Time Frame: Parts 2 and 4: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: PK Set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in the urine. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 4: MRD: TAK-041 160/80 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 15
ng/mL | 549.7 (146.05) | 879.7 (217.95) | 1260.8 (265.22) | 1760.0 (349.69) | 1266.5 (366.10)

12. Secondary Outcome: Part 1: Tmax: Time to Reach the Cmax for TAK-041 in SRD Participants [Day 1]
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hours | 0.992 [0.48 to 3.00] | 1.742 [1.03 to 2.00] | 3.000 [1.00 to 48.02] | 13.017 [1.50 to 96.05] | 13.517 [1.98 to 71.97]

13. Secondary Outcome: Part 1: Tmax: Time to Reach the Cmax for TAK-041 in SRD Participants [Day 8], Cohorts 1 (20 mg) and 2 (40 mg) Only
Time Frame: Part 1: Pre-dose on Day 8 and at multiple timepoints (Up to 96 hours) post-dose
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg
Number analyzed (Participants) | 6 | 6
hours | 1.992 [1.00 to 3.00] | 1.583 [1.50 to 2.00]

14. Secondary Outcome: Parts 2 and 4: Tmax: Time to Reach the Cmax for TAK-041 in MRD Participants [Day 1]
Time Frame: Parts 2 and 4: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 4: MRD: TAK-041 160/80 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 15
hours | 2.517 [0.97 to 4.00] | 1.525 [1.50 to 3.05] | 2.500 [1.50 to 47.88] | 3.000 [1.50 to 95.77] | 2.000 [1.00 to 96.80]

15. Secondary Outcome: Part 3: Tmax: Time to Reach the Cmax for TAK-041 in RBA/Food Effect Participants [Day 1]
Time Frame: Part 3: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part3:RBA/Food Effect:Regimen C-Part 1 Cohort2,Part 2 Cohort 1
Number analyzed (Participants) | 9 | 9 | 12
hours | 2.000 [0.98 to 36.00] | 2.000 [2.00 to 23.92] | 1.817 [0.97 to 4.00]

16. Secondary Outcome: Part 1: AUC24: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-041 in SRD Participants [Day 1]
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL | 1662.3 (390.74) | 2844.6 (263.78) | 15594.9 (5560.51) | 22471.2 (4340.25) | 21426.6 (6026.07)

17. Secondary Outcome: Part 1: AUC24: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-041 in SRD Participants [Day 8], Cohorts 1 (20 mg) and 2 (40 mg) Only
Time Frame: Part 1: Pre-dose on Day 8 and at multiple timepoints (Up to 96 hours) post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg
Number analyzed (Participants) | 6 | 6
h*ng/mL | 6399.5 (1809.44) | 11955.2 (1091.59)

18. Secondary Outcome: Parts 2 and 4: AUC24: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-041 in MRD Participants [Day 1]
Time Frame: Parts 2 and 4: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 4: MRD: TAK-041 160/80 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 15
h*ng/mL | 9188.0 (3095.87) | 14556.7 (4317.73) | 22450.3 (3625.16) | 28014.6 (7698.01) | 20400.8 (5096.46)

19. Secondary Outcome: Part 3: AUC24: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours for TAK-041 in RBA/Food Effect Participants [Day 1]
Time Frame: Part 3: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part3:RBA/Food Effect:Regimen C-Part 1 Cohort2,Part 2 Cohort 1
Number analyzed (Participants) | 9 | 9 | 12
h*ng/mL | 11940.8 (3052.59) | 13827.9 (5143.36) | 10571.6 (2643.23)

20. Secondary Outcome: Part 1: AUC96: Area Under the Plasma Concentration-Time Curve From Time 0 to 96 Hours for TAK-041 in SRD Participants [Day 1]
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL | 5237.2 (1107.97) | 9746.9 (781.89) | 59514.3 (14414.25) | 92784.6 (13410.06) | 90585.1 (15742.96)

21. Secondary Outcome: Part 1: AUC96: Area Under the Plasma Concentration-Time Curve From Time 0 to 96 Hours for TAK-041 in SRD Participants [Day 8], Cohorts 1 (20 mg) and 2 (40 mg) Only
Time Frame: Part 1: Pre-dose on Day 8 and at multiple timepoints (Up to 96 hours) post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg
Number analyzed (Participants) | 6 | 6
h*ng/mL | 21180.0 (5680.75) | 40487.8 (3088.81)

22. Secondary Outcome: Parts 2 and 4: AUC96: Area Under the Plasma Concentration-Time Curve From Time 0 to 96 Hours for TAK-041 in MRD Participants [Day 1]
Time Frame: Parts 2 and 4: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 4: MRD: TAK-041 160/80 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 15
h*ng/mL | 35102.6 (6612.50) | 60770.4 (15609.67) | 91712.9 (12328.54) | 123645.0 (29616.79) | 90372.3 (22678.03)

23. Secondary Outcome: Part 1: AUCt: Area Under the Plasma Concentration-Time Curve From Time 0 to Time t for TAK-041 in SRD Participants [Day 1]
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL | 18038.1 (9735.91) | 44649.4 (5067.39) | 251124.1 (67210.68) | 344075.1 (145462.41) | 361251.2 (97096.24)

24. Secondary Outcome: Part 1: AUCt: Area Under the Plasma Concentration-Time Curve From Time 0 to Time t for TAK-041 in SRD Participants [Day 8], Cohorts 1 (20 mg) and 2 (40 mg) Only
Time Frame: Part 1: Pre-dose on Day 8 and at multiple timepoints (Up to 96 hours) post-dose
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg
Number analyzed (Participants) | 6 | 6
h*ng/mL | 104692.7 (48397.26) | 202185.0 (38724.05)

25. Secondary Outcome: Parts 2 and 4: AUCt: Area Under the Plasma Concentration-Time Curve From Time 0 to Time t for TAK-041 in MRD Participants [Day 1]
Time Frame: Parts 2 and 4: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 4: MRD: TAK-041 160/80 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 15
h*ng/mL | 55530.5 (7016.30) | 99401.9 (25287.60) | 147300.0 (16846.42) | 203506.2 (49784.48) | 148889.0 (40389.92)

26. Secondary Outcome: Part 3: AUCt: Area Under the Plasma Concentration-Time Curve From Time 0 to Time t for TAK-041 in RBA/Food Effect Participants [Day 1]
Time Frame: Part 3: Day 1 pre-dose and at multiple time points (up to 96 hours) post-dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part3:RBA/Food Effect:Regimen C-Part 1 Cohort2,Part 2 Cohort 1
Number analyzed (Participants) | 9 | 9 | 12
h*ng/mL | 116064.6 (36590.93) | 126001.0 (34652.19) | 128857.7 (81053.57)

27. Secondary Outcome: Part 1: AUCinf: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for TAK-041 in SRD Participants [Day 1]
Time Frame: as for outcome 9
Population: PK Set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in the urine. For Part 1 (SRD): Cohorts 1 and 2: TAK-041 5 and 10 mg respectively data could not be analyzed as follow-up time was not enough to calculate AUC0-inf because of the long half-life of TAK-041.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg
Number analyzed (Participants) | 0 | 0 | 6 | 6 | 6
h*ng/mL |  |  | 283461.1 (96704.07) | 381403.3 (208693.96) | 395932.4 (129676.19)

28. Secondary Outcome: Part 1: AUCinf: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for TAK-041 in SRD Participants [Day 8], Cohorts 1 (20 mg) and 2 (40 mg) Only
Time Frame: Part 1: Pre-dose on Day 8 and at multiple timepoints (Up to 96 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg
Number analyzed (Participants) | 4 | 6
h*ng/mL | 122801.1 (40764.68) | 203288.4 (39395.16)

29. Secondary Outcome: Parts 2 and 4: AUCtau: Area Under the Plasma Concentration-Time Curve From Time 0 to Time Tau Over the Dosing Interval for TAK-041 in MRD Participants [Day 1]
Time Frame: Parts 2 and 4: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 4: MRD: TAK-041 160/80 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 15
h*ng/mL | 55530.5 (7016.30) | 99401.9 (25287.60) | 147300.0 (16846.42) | 203506.2 (49784.48) | 148889.0 (40389.92)

30. Secondary Outcome: Part 1: T1/2z: Terminal Disposition Phase Half-Life for TAK-041 in SRD Participants [Day 1]
Time Frame: as for outcome 9
Population: PK Set included all participants who received study drug and had at least 1 measurable plasma concentration or amount of drug in the urine. For Part 1 (SRD): Cohorts 1 and 2: TAK-041 5 and 10 mg respectively data could not be analyzed as follow-up time was not enough to calculate T1/2z because of the long half-life of TAK-041.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg
Number analyzed (Participants) | 0 | 0 | 6 | 6 | 6
hours |  |  | 284.0 [107 to 431] | 208.0 [55 to 450] | 260.6 [108 to 402]

31. Secondary Outcome: Part 1: T1/2z: Terminal Disposition Phase Half-Life for TAK-041 in SRD Participants [Day 8], Cohorts 1 (20 mg) and 2 (40 mg) Only
Time Frame: Part 1: Pre-dose on Day 8 and at multiple timepoints (Up to 96 hours) post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg
Number analyzed (Participants) | 4 | 6
hours | 312.4 [185 to 367] | 306.3 [197 to 405]

32. Secondary Outcome: Parts 2 and 4: T1/2z: Terminal Disposition Phase Half-Life for TAK-041 in MRD Participants [Day 1]
Time Frame: Parts 2 and 4: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 4: MRD: TAK-041 160/80 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 13
hours | 196.2 [61 to 891] | 313.1 [158 to 376] | 153.5 [97 to 273] | 263.0 [96 to 420] | 300.1 [145 to 572]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 42 days after the last dose of study drug (Up to 12 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1 (SRD): Placebo Cohorts 1-5 | Part 1 (SRD): Cohort 1: TAK-041 5 mg | Part 1 (SRD): Cohort 2: TAK-041 10 mg | Part 1 (SRD): Cohort 1: TAK-041 20 mg | Part 1 (SRD): Cohort 2: TAK-041 40 mg | Part 1 (SRD): Cohort 3: TAK-041 80 mg | Part 1 (SRD): Cohort 4: TAK-041 120 mg | Part 1 (SRD): Cohort 5: TAK-041 160 mg | Part 2 (MRD): Placebo Cohorts 1-4 | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A | Part 3: RBA/Food Effect: Regimen B | Part 4: MRD: Placebo | Part 4: MRD: TAK-041 160/80 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/8 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/8 | 0/16
Other Adverse Events (participants affected / at risk) | 4/10 | 0/6 | 0/6 | 0/6 | 0/6 | 2/6 | 2/6 | 2/6 | 3/8 | 4/6 | 4/6 | 3/6 | 5/6 | 1/9 | 2/9 | 6/8 | 9/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 (SRD): Placebo Cohorts 1-5 (N=10) | Part 1 (SRD): Cohort 1: TAK-041 5 mg (N=6) | Part 1 (SRD): Cohort 2: TAK-041 10 mg (N=6) | Part 1 (SRD): Cohort 1: TAK-041 20 mg (N=6) | Part 1 (SRD): Cohort 2: TAK-041 40 mg (N=6) | Part 1 (SRD): Cohort 3: TAK-041 80 mg (N=6) | Part 1 (SRD): Cohort 4: TAK-041 120 mg (N=6) | Part 1 (SRD): Cohort 5: TAK-041 160 mg (N=6) | Part 2 (MRD): Placebo Cohorts 1-4 (N=8) | Part 2 (MRD): Cohort 1: TAK-041 40/20 mg (N=6) | Part 2 (MRD): Cohort 2: TAK-041 80/40 mg (N=6) | Part 2 (MRD): Cohort 3: TAK-041 120/60 mg (N=6) | Part 2 (MRD): Cohort 4: TAK-041 160/80 mg (N=6) | Part 3: Relative Bioavailability (RBA)/Food Effect: Regimen A (N=9) | Part 3: RBA/Food Effect: Regimen B (N=9) | Part 4: MRD: Placebo (N=8) | Part 4: MRD: TAK-041 160/80 mg (N=16)
Application site dermatitis (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site phlebitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Energy increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Change in sustained attention (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT02748694/SAP_000.pdf
  • Study Protocol (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT02748694/Prot_001.pdf